# STATISTICAL ANALYSIS PLAN

#### LT4090-201

A phase II, multicenter, randomized, investigator-masked, 3-parallel groups study to evaluate efficacy and safety of T4090 ophthalmic solution (preservative-free Kinezodianone R HCl 0.2% or 0.3%) versus Rhopressa® ophthalmic solution (preserved netarsudil 0.02%) in patients with open-angle glaucoma or ocular hypertension

AUTHOR:

VERSION NUMBER AND DATE: V2.0, 06JAN2025

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_\V2.0

Author: Version Number: 2.0



## STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan V2.0 (Dated 06JAN2025) for Protocol LT4090-201.

| | Name | Signature | Date |
|-----------|-----------------------|---------------------|------|
| Author: | | Refer to eSignature | |
| Position: | Statistical Team Lead | | |
| Сотрапу: | | | |

Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.

| | Name | Signature | Date |
|--------------|------------------------------|---------------------|------|
| Approved By: | | Refer to eSignature | |
| Position: | Senior Biostatistical Review | er | |
| Company: | | | |
| | • | | |
| Approved By: | | Refer to eSignature | |
| Position: | Medical Development Direct | tor | |
| Company: | Laboratoires Théa | | |
| Approved By: | | Refer to eSignature | |
| Position: | Biometrics Manager | ' | |
| Сотрапу: | Laboratoires Théa | | |

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_\V2.0


# TABLE OF CONTENTS

| 1. | INTRODUCTION | | 15 |
|---|---|---|---|
| 2. | STUDY OBJECTIVES AND ESTIMANDS | | 15 |
| 2.1. | Primary Objective | | 15 |
| 2.3. | Estimands | | 15 |
| 3. | STUDY DESIGN | | 19 |
| 3.1. | General Description | | 19 |
| 3.2. | Sample Size | | 21 |
| 3.3. | Schedule of Events | | 21 |
| 3.4. | Changes to Analysis from Protocol | | 21 |
| 4. | PLANNED ANALYSES | | 23 |
| 4.1. | Data Monitoring Committee (DMC) | | 23 |
| 4.2. | Interim Analysis | | 23 |
| 4.3. | Final Analysis | | 23 |
| 5. | ANALYSIS SETS | | 23 |
| 5.1. | All Patients Screened Set [SCR] | | 23 |
| 5.2. | Intent-to-Treat Set [ITT] | | 23 |
| 5.3. | Full Analysis Set [FAS] | | 24 |
| 5.4. | Per-Protocol Analysis Set [PP] | | 24 |
| 5.5. | Safety Analysis Set [SAF] | | 25 |
| Docu | ment:\Biostatistics\Documentation\SAP\ T4090-201_Statistica | l Analysis Plan_∀2.0 | |
| Autho | or: | Version Number: | 2.0 |
| | | Version Date: | 06JAN2025 |

# Statistical Analysis Plan 6. GENERAL CONSIDERATIONS ......25 6.1. 6.2. 6.7. 6.8. 7. **7.1.** 7.3. 7.5. 8. 9. 9.1. 9.2. Document: ...\Biostatistics\Documentation\SAP\ T4090-201 Statistical Analysis Plan V2.0 Version Number: Author: 2.0 Version Date: 06JAN2025

2.0

06JAN2025



Statistical Analysis Plan

Author:

| 10. | DEMO | OGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 34 |
|---|---|---|---|
| 11. | HISTO | ORY OF GLAUCOMA OR OHT | 35 |
| 12. | MEDI | CAL AND SURGICAL HISTORY AND CURRENT CONDITIONS | 36 |
| 13. | MEDI | CATIONS | 37 |
| 14. | STUD | Y TREATMENT EXPOSURE | 37 |
| 15. | STUD | Y TREATMENT COMPLIANCE | 38 |
| 16. | EFFIC | CACY OUTCOMES | 38 |
| 16.1.<br>16.1<br>16.1 | | mary Efficacy mary Efficacy Endpoint & Derivation | |
| Docum | ent: | \Riostatistics\Documentation\SAP\ T4090-201 Statistical Analysis Plan \/2 0 | |

Version Number:

Version Date:





## LIST OF ABBREVIATIONS

| Abbreviation | Term |
|--------------|-----------------------------------------|
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ATC | Anatomical Therapeutic Chemical |
| CEC | Corneal Endothelial Cells |
| CI | Confident Interval |
| eCRF | Electronic Case Report Form |
| ICH | International Council for Harmonization |
| IMP | Investigational Medicinal Product |
| IOP | Intra-Ocular Pressure |
| IRT | Interactive Response Technology |
| ITT | Intent-To-Treat |

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_\V2.0


| Abbreviation | Тегт |
|--------------|----------------------------------------------|
| LS | Least Squares |
| MDC | Multiple-Dose Container |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MH | Medical History |
| MMRM | Mixed Model for Repeated Measures |
| NA | Not Applicable |
| OAG | Open-Angle Glaucoma |
| OHT | Ocular Hypertension |
| PD | Protocol Deviation |
| PF | Preservative-Free |
| PP | Per-Protocol |
| PT | Preferred Term |
| REML | Restricted Maximum Likelihood |

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_\V2.0


| Abbreviation | Term |
|--------------|-----------------------------------------------|
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Standard Deviation |
| SDC | Single-Dose Container |
| SE | Standard Error |
| SOC | System Organ Class |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TEAE | Treatment Emergent Adverse Event |
| UD | Unit Dose |
| WHO-DD | World Health Organization Drug Dictionary |

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V2.0




### 1. Introduction

This statistical analysis plan (SAP) describes the rules and conventions to be used in the presentation and analysis of efficacy and safety data for Protocol LT4090-201. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This SAP is based on Protocol version 2.0 dated 17 April 2024, Protocol Clarification Letter #1 dated 10 June 2024, Protocol Clarification Letter #2 dated 10 July 2024, and electronic Case Report Form (eCRF) version 3.0 dated 27 September 2024.

#### 2. STUDY OBJECTIVES AND ESTIMANDS

### 2.1. Primary Objective

The primary objective of the study is to compare the ocular hypotensive efficacy of two concentrations of T4090 (Kinezodianone R HCl 0.2 % and 0.3 %) ophthalmic solution with Rhopressa® ophthalmic solution.

#### 2.3. Estimands

The primary, and secondary estimands to support regulatory decisions are described in the following table:

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_\V2.0


### Table A Objectives and Estimands

### Primary Efficacy:

| | | | Attributes | | |
|---|---|---|---|---|---|
| Objective | Estimands | Treatment | Population | Variable/<br>Endpoint | Population-Level Summary<br>Measure |
| To compare the ocular hypotensive efficacy of two concentrations of T4090 (Kinezodianone R HCl 0.2 % and 0.3 %) ophthalmic solution with Rhopressa® ophthalmic solution, and to compare T4090 0.2% with T4090 0.3% | Primary<br>Estimand | T4090 0.2 % or T4090 0.3% or Rhopressa® (administered once daily in each eye) | Patients in whom both eyes were diagnosed with ocular hypertension (OHT) or openangle glaucoma (OAG), and further defined through the inclusion and exclusion criteria | Change from<br>baseline in<br>the mean<br>diurnal intra-<br>ocular<br>pressure<br>(IOP) at<br>Week 7 in the<br>study eye* | Least squares (LS) means of change from baseline in mean diurnal IOP at Week 7 based on a mixed model with repeated measures (MMRM), with test of treatments effect based on differences of LS means. |

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0

Author: Version Number: 1.0

#### 3. STUDY DESIGN

### 3.1. General Description

This is a phase II, multicenter, randomized, investigator-masked, 3-parallel groups, 7-week treatment duration in patients with OAG or OHT. Approximately 126 eligible patients (naïve or using ocular hypotensive medication) were planned to be randomized on a 1:1:1 basis to T4090 (PF Kinezodianone R HCl 0.2% or 0.3%) or Rhopressa®.

The randomization lists are generated using a validated system, which involves a pseudo-random number generator so that the resulting sequence of treatments will be both reproducible and non-predictable. Access to the codes will be controlled and documented.

Randomized patients will attend 3 visits (Visit #3 to #5) at the investigator center during the study treatment period:

- Visit #1: Screening visit,
- Visit #1.1: Optional visit planned according to the investigator's judgement,
- Visit #1.2: Visit in case of extension of the washout period,
- Visit #2 Day 1 (D1): Randomization visit,
- Visit #3 Week 2 (W2) Day 15 (±2 days),
- Visit #4 Week 4 (W4) Day 29 (±3 days),
- Visit #5 Week 7 (W7) Day 50 (±3 days): End of treatment visit.

At the Randomization visit (D1; Visit #2), patients will be randomly assigned, after stratification according to their baseline IOP at 8:00 AM to one of the following 3 treatment arms:

#### Test product:

- T4090 (PF Kinezodianone R HCl 0.2%) ophthalmic solution, in single-dose container (SDC),
- T4090 (PF Kinezodianone R HCl 0.3%) ophthalmic solution, in SDC.

#### Reference product:

Rhopressa® (preserved netarsudil 0.02%) ophthalmic solution, in multiple-dose container (MDC).

The patient will administer the assigned treatment (T4090 0.2% or T4090 0.3% or Rhopressa®) once daily at 8:00 PM (±1 hour) in the conjunctival cul-de-sac of each eye from Day 1 to the day before the End of treatment visit (Week 7; Visit #5).

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0


Version Date: 13Nov2024

The maximum study duration will be 12 weeks: 5-week washout period (including optional 1-week washout extension) (See Section 3.1.1 of the Protocol), and 7-week treatment period. A minimum of 4 visits and a maximum of 7 visits are planned. The number of visits will depend on the patient's screening status (naïve patient or patient using ocular hypotensive medication).

Figure A Overall design of the study (pre-treated patient)



Figure B Overall design of the study (naïve patient)



Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0


## 3.2. Sample Size

This is a Phase II pilot study, and the analysis is to be considered as exploratory. Therefore, no formal sample size calculation is performed. It is planned to randomize 126 patients with a randomization scheme 1:1:1 with a stratification by baseline IOP at 8:00 AM in class

### 3.3. Schedule of Events

Schedule of events can be found in Section 6.1 of the Protocol.

| 3.4. | Changes | to A | analysis | from | Proto | col |
|------|---------|------|----------|------|-------|-----|
|------|---------|------|----------|------|-------|-----|

| provi<br>categ<br>will t | e protocol S<br>ided for cor<br>gorical varia<br>be displayed<br>ssary. | itinuous v<br>ibles.". T | variables<br>his has b | s and 95%<br>been upd | % CI of tated in S | the propo<br>Section 8 | rtion wil | ll be displ<br>AP to ex | layed for | each mo | odality o<br>f the pro |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | d for each | ı modali | ty of cate | egorical | variables | s", as CI | for categ | orical va | riables v | was not d |
| ument: | \Biostat | tistics\Do | cumenta | ation\SAF | P\ T4090 | 0-201_Sta | | analysis P | _ | | |

| Statistical Analysis Plan | |
|---|---|
| <u> </u> | |
| † | |
| _ | MMRM model "will include treatment, visit (W2, W4 |
| and W7), baseline mean diurnal IOP, baseline IOF | out 8:00 AM in class |
| | Section 16.1.3 of this SAP to exclude "baseline IOP at |
| _ | to potential collinearity. In addition, "and patient ID as |
| | ation purposes, as no separate random statement with |
| patient ID is required in the analysis model. | |
| _ | |
| - | |
| • | |
| Document:\Biostatistics\Documentation\SAP\ T4090 | -201 Statistical Analysis Plan V1.0 |

#### 4. PLANNED ANALYSES

The following analysis will be performed for this study:

Final analysis

### 4.1. Data Monitoring Committee (DMC)

There will be no DMC for this study.

### 4.2. Interim Analysis

There will be no interim analysis for this study.

### 4.3. Final Analysis

All final, planned analyses identified in this SAP will be performed by following Customer

Authorization of this SAP, Database Lock, Customer Authorization of Analysis Sets and Unblinding of Treatment.

### 5. ANALYSIS SETS

The following analysis sets will be considered.

Agreement and authorization of patients included/excluded from each analysis set will be conducted prior to the unblinding of the study.

# 5.1. All Patients Screened Set [SCR]

The all patients screened (SCR) set will contain all patients who provide informed consent for this study.

# 5.2. Intent-to-Treat Set [ITT]

The intent-to-treat (ITT) set will contain all patients who were randomized. For analyses and displays based on ITT, patients will be classified according to randomized treatment.

| Document: | \Biostatistics\Documentation\SAP\ T4090 | 0-201_Statistical Analysis Plan_V1.0 |
|---|---|---|

#### **5.3. Full Analysis Set [FAS]**

The full analysis set (FAS) will contain all patients in the ITT set who received at least one dose of study treatment. For analyses and displays based on FAS, patients will be classified according to randomized treatment.

The FAS will be the primary population for efficacy analysis.

| 5.4. | Per-Protocol Analysis Set [PP] | |
|---|---|---|
| The perexclusio | -protocol (PP) analysis set will contain all patients in the FAS who did not | experience any reason for |
| Toward of the state of the stat | | |
| | lyses and displays based on PP set, patients will be classified according to set will be considered as secondary population | reatment received. |
| Docume<br>Author: | Versio | s Plan_V1.0<br>n Number: 1.0<br>n Date: 13Nov2024 |

### 5.5. Safety Analysis Set [SAF]

The safety (SAF) analysis set will contain all patients who received at least one dose of study treatment. For analyses and displays based on SAF, patients will be classified according to treatment received.

The safety set will be the primary population for safety analysis.

### **6. GENERAL CONSIDERATIONS**

### **6.1.** Reference Start Date and Study Day

Reference start date is defined as the day of the first dose of study treatment (Day 1 is the day of the first dose of study treatment).

Study day will be calculated from the reference start date and will be used to show start/end day of assessments and events. It will appear in every listing where an assessment date or event date appears.

- If the date of the event is on or after the reference date, then: Study Day = (date of event – reference date) + 1.
- If the date of the event is prior to the reference date, then: Study Day = (date of event – reference date).

In the situation where the event date is partial or missing, the date, study day, and any corresponding durations will appear partial or missing in the listings.

#### 6.2. Baseline

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to or on date of first dose of study treatment, excluding measurements reported during washout period (i.e., from Screening visit through to the day prior to Randomization visit) for pre-treated patients. No imputation will be performed if baseline measurement is missing.

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0


| Statistical Ana | alysis Plan | | | | |
|---|---|---|---|---|---|
| value recorded a | | mization visit, r | espectively at 10 | 0:00 AM and at 4:00 PM | diurnal IOP. For IOP, the<br>M, will be the baseline |
| | | <del></del> | | | |
| Document: | .\Biostatistics\Docun | nentation\SAP\ 1 | Γ4090-201_Stati | stical Analysis Plan_V1 | 1.0 |
| Author: | | | | Version Number | |

| | | DL LT4090-201 |
|---|---|---|
| Statistical Analysis Plan | | |
| | | • |
| 6.7. Statistical Tests | | |
| The default significant level will be 5% and no adjustment of the | type I error rate will be | |
| will be 95% and all tests will be two-sided, unless otherwise spec | | dence intervals<br>yses. |
| For continuous quantitative parameters, treatment groups will be | compared using an MMRM. | |
| Document:\Biostatistics\Documentation\SAP\ T4090-201_S | Statistical Analysis Plan V1.0 | |

#### 6.8. Common Calculations

For quantitative measurements, absolute and percent change from baseline will be calculated as:

- Absolute change = Test Value at Visit X Baseline Value,
- Percent change = (Absolute change / Baseline Value) \*100.

### 7. STATISTICAL CONSIDERATIONS

## 7.1. Adjustments for Covariates and Factors to be Included in Analyses

The following covariates and factors will be used in the analyses. For details of their inclusion in the models, see the specific analysis section.

- Baseline IOP continuous value,
- Treatment (T4090 0.2%, T4090 0.3%, and Rhopressa®),
- Visit (W2, W4, and W7).

# 7.3. Missing Data

Missing safety data will not be imputed unless described in the specific analysis section. Missing efficacy data will be handled as described in Section 16 of this SAP.

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0


| Statistical Analysis Plan | | |
|---|---|---|
| TE M Wale Commenter of M Walland | | |
| 7.5. Multiple Comparisons/ Multiplicity | | |
| Analysis will be performed to common officers and sinte between the | ant groups (and T4000 | aanaantrati |
| Analyses will be performed to compare efficacy endpoints between treatn | | |
| versus Rhopressa® and both T4090 concentrations comparison). All analy | ses are considered as sup | portive and any |
| Document:\Biostatistics\Documentation\SAP\ T4090-201_Statistical | Analysis Plan_V1.0 | |



statistical test comparing treatment groups will be made without adjustment for multiplicity.

### 8. OUTPUT PRESENTATIONS

Variables recorded for each eye will be described separately for the study eye and for the contralateral eye (if applicable).

Continuous variables will be summarized using descriptive statistics: number of non-missing observations (n), mean, standard deviation (SD), median, lower quartile (Q1), upper quartile (Q3), minimum (Min) and maximum (Max). When applicable, 95% confidence interval (CI) of the mean will be provided for continuous variables.

Categorical variables will be summarized using frequency distribution: number of non-missing observations (n), count and percentages (%, based on n unless otherwise indicated in the table template) of each modality.

### 9. DISPOSITION AND WITHDRAWALS

All patients who provided informed consent will be accounted for in this study.

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0


### 9.1. Disposition

Patient disposition and withdrawals, including number of patients screened/randomized and reasons of discontinued treatment or study, will be presented for the SCR set.

A listing of all disposition data, including early treatment and study discontinued patients and reasons of withdrawals, will be provided for the SCR set.

Details of any inclusion/exclusion criteria which were not met will be listed for the SCR set, including the protocol version(s) under which each patient was consented.

The number (%) of patients included in each analysis set (ITT, FAS, PP and SAF) and reason for exclusion from each analysis set will be presented by treatment group and overall, for the ITT set.

A listing of patients with analysis sets inclusion and the reason for exclusion from ITT, FAS, PP and SAF, and including treatment group (planned group and actual group), will be produced for the SCR set.

#### 9.2. Protocol Deviations

The number (%) of patients with deviations by PD category will be presented in a summary table by treatment group and overall for the ITT set, including:

- Patients with at least one PD
- Patients with at least one critical PD
- Patients with at least one major PD
- Patients with at least one minor PD
- Patients with at least one important PD

A listing of all PDs will be provided for the ITT set.

#### 10. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic data and other baseline characteristics will be presented by treatment group and overall for the FAS,

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0


| Statistical Analysis Plan | | |
|---|---|---|
| and for PP and SAF sets demographic or other baseline characteristics. The following demograph reported for this study: | No statistical testing will be carried out hic and other baseline characteristics wi | |
| Demographics: | | |
| <ul> <li>Age (years) – as continuous, and in two classes: Adult (18-64), 0</li> <li>Sex (Male, Female),</li> <li>Race (American Indian or Alaska Native, Asian, Black or Africa Pacific Islander, White, Not Reported, Unknown),</li> <li>Ethnicity (Hispanic or Latino, Not Hispanic or Latino, Not Reported (Blue, Gray, Green, Brown, Hazel, Other),</li> <li>Baseline IOP at 8:00 am in the study eye in classes</li> </ul> | an American, Native Hawaiian or Other | : |
| A listing of the above demographic data will be provided for the FAS. T | This listing will also include: | |
| <ul> <li>Childbearing potential (Yes, No) and birth control method – for</li> <li>Study Eye (Right, Left), as determined in Section 6.6.</li> </ul> Baseline values of the efficacy and safety endpoints will be provided in standard W4, and W7. | | 2, |
| 11. HISTORY OF GLAUCOMA OR OHT | | |
| History of glaucoma or OHT presented for the FAS, and for PP and SAF sets variables will be summarized by treatment group and overall: • Treatment status (Naive patient, Previously treated patient), • Type of previous antiglaucoma treatment (if applicable) • For each eye: | will . The following | be |
| Document:\Biostatistics\Documentation\SAP\ T4090-201_Statistica | cal Analysis Plan_V1.0 | |
| Author: | Version Number: Version Date: 13Nov26 | 1.0<br>024 |





# 13. MEDICATIONS

| Medications reported treatment group, for the FAS, and for PP and SAF sets | will be summarized overall and | by |
|---|---|---|
| Medications will be coded using World Health Organization-Drug Diction higher. | ary (WHO-DD) Version March 2024 | or |
| Medication will be presented by Anatomical Therapeutic Chemical (ATC) | Level 2 and Level 4. Separate summaries for pr | rior |
| and concomitant medications based on ocular location (Ocular vs Systemic | • | .101 |
| A listing for all prior and concomitant medications will be provided for the | e FAS. | |
| 14. STUDY TREATMENT EXPOSURE | | |
| Exposure to study treatment in days will be presented by treatment group | for the SAF set. | |
| Document:\Biostatistics\Documentation\SAP\ T4090-201_Statistical Author: | _ | 1.0 |
| | Version Date: 13Nov20 | |

### 15. STUDY TREATMENT COMPLIANCE

| _ | |
|---|---|
| _ | • |

Compliance (%) to study treatment will be presented separately for the study eye and the contralateral eye by treatment group for the SAF set.

Listings of all data related to study treatment administration, including interruptions, missed doses and time modifications, exposure and compliance will be provided for the SAF set.



# 16. EFFICACY OUTCOMES

# 16.1. Primary Efficacy

For this study, the primary clinical question of interest is to compare the ocular hypotensive efficacy of two concentrations of T4090 ophthalmic solution with Rhopressa® ophthalmic solution in terms of lowering the mean diurnal IOP at Week 7 in the study eye (see Section 6.6).

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0




Document:

Author:

### 16.1.1. Primary Efficacy Endpoint & Derivation

The primary efficacy endpoint is the change from baseline (see calculation in Section 6.8) in the mean diurnal IOP at Week 7 in the study eye.

Mean diurnal IOP\* = (IOP at 8:00 AM + IOP at 10:00 AM + IOP at 4:00 PM) / 3 \* If IOP value is missing at any timepoint, the mean diurnal IOP will be missing.

Version Number:

Version Date:

1.0

13Nov2024

...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0



#### 16.1.3. Primary Analysis of Primary Efficacy Endpoint (Primary Estimand)

Descriptive statistics for mean diurnal IOP and change from baseline at Week 7 in the study eye will be provided by treatment group on the FAS.

The primary objective of this study is to test the hypothesis (H0) that there is no difference in change from baseline in the mean diurnal IOP at Week 7 among treatment groups. H0 will be tested against the alternative hypothesis H1 of at least one of the test groups is different to reference group at 0.05 alpha level.

The primary efficacy analysis, performed for the FAS, is evaluated using a restricted maximum likelihood (REML) based, mixed-effects model for repeated measures (MMRM) estimating change from baseline across post-baseline visits. The model will include the fixed, categorical effects of treatment (T4090 0.2%, T4090 0.3%, and Rhopressa®), visit (W2, W4, and W7), and treatment-by-visit interaction, as well as the fixed, continuous covariates of baseline mean diurnal IOP value and baseline value-by-visit interaction (see Section 7.1). The general form of the model will then be:

Change = Baseline + Treatment + Visit + Treatment\*Visit + Baseline\*Visit



Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0






Separate descriptions of treatment-emergent ocular and systemic TEAEs will be performed by treatment group:

- Number and percentage of patients experiencing at least one TEAE, serious TEAE, study treatment related
  TEAE, study treatment related serious TEAE, TEAE leading to study treatment discontinuation, TEAE
  leading to death, TEAE by maximum severity, and treatment-emergent adverse event of special interest
  (AESI only for ocular AEs),
- Number and percentage of patients experiencing at least one TEAE, as well as the number of TEAEs, by SOC and PT. The same summary table will be performed for serious TEAEs, study treatment related TEAEs, study treatment related serious TEAEs, TEAEs leading to study treatment discontinuation, and treatment-emergent AESI (only ocular),
- Number and percentage of patients experiencing at least one TEAE, by SOC, PT, and maximum severity.
   The same summary table will be performed for study treatment related TEAEs,
- Number and percentage of patients experiencing at least one TEAE, by SOC, PT, and maximum relationship
  to study treatment.

| Listings will include all AEs (TEAEs and non-TI | EAEs) |
|-------------------------------------------------|-------|
|-------------------------------------------------|-------|

#### **17.1.1.** All TEAEs

Incidence of TEAEs will be presented by SOC and PT and broken down further by maximum severity and maximum relationship to study treatment.

#### 17.1.1.1. SEVERITY

Severity is classed as "mild", "moderate", and "severe" (increasing severity).

If a subject reports a TEAE more than once within that SOC/ PT, the AE with the highest severity will be used in the corresponding severity summaries.

#### 17.1.1.2. RELATIONSHIP TO STUDY TREATMENT

Relationship, as indicated by the masked investigator, is classed as "not related", and "related" (increasing severity of relationship).

If a subject reports the same AE more than once within that SOC/ PT, the AE with the worst-case relationship to study treatment will be used in the corresponding relationship summaries.

| study detailment will be used in the corresponding re- | actionship summaries. | |
|---|---|---|
| ocument:\Biostatistics\Documentation\SAP\ T4090-201_Statistical Analysis Plan_V1.0 | | |
| | Version Number: | 1.0 |
| | , , , | Version Number: |

#### 17.1.2. TEAEs Leading to Discontinuation of Study Treatment

A summary of TEAEs leading to

discontinuation of study treatment by SOC and PT will be prepared.

#### 17.1.3. Serious Adverse Events

A summary of

serious TEAEs by SOC and PT will be prepared.

#### 17.1.4. Adverse Events Leading to Death

The number of patients with TEAEs leading to death will be included in the overview TEAE summary table. The summary by SOC and PT will be part of the serious TEAE summary.

#### 17.1.5. Adverse Events of Special Interest

Based on observations from previous studies with ROCKi, the following AEs will be considered as AESI, if judged significant by the investigator:

- All AEs related to CEC
- All AEs related to visual impairment (partial or total visual acuity loss)
- Corneal opacity
- Lens opacity/cataract
- Corneal verticillate

A summary of treatment-emergent (ocular) AESIs by SOC and PT will be prepared.

#### **17.2.** Deaths

If any subject dies during the study the study that it is a data listing.

Document: ...\Biostatistics\Documentation\SAP\ T4090-201\_Statistical Analysis Plan\_V1.0
